CLINICAL TRIAL: NCT05708651
Title: Tematic Evaluation of a New Medical Device (STAIRWAY) for Open Airways
Brief Title: Evaluation of Medical Device for Airway Patency During Sedation (SW01-2022)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stairway Medical AB (Industry)
Collaborators: Lund University (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIV-22-09-040787; Dnr: 5.1-2022-75020 (Other: Medical Products Agency (Sweden))
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Airway Obstruction; Sedation Complication; Safety Issues; Patient Satisfaction; Work Related Stress; Breathing Arrested; Complication of Treatment; Hypoxia
Keywords: Sedation, procedural; Airway patency; Device, medical; Patient safety; Respiratory depression; Breathing, spontaneous; Propofol; Sedation, level; Biteblock
MeSH Terms: conditions — Airway Obstruction; Patient Satisfaction; Occupational Stress; Apnea; Hypoxia; Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Four-part preclinical [I-II] and clinical [III-IV] trial carried out, in 12 + 12 volunteer study participants [I-II] and in 16 + 16 study patients [III-IV)], according to an intra-individual randomised paired crossover study design, where the investigational device is compared with standard procedure (comparator; biteblock [I-II] or no device [II-IV]) for airway patency (tidal volume [I], transpharyngeal distance [II], signs of airway obstruction [III-IV], use of manual airway support [III-IV]).
Who Masked: Outcomes Assessor
Masking Description: All study data recorded on-site will be masked for investigational device or comparator (and recorded in individually randomized order) in the study protocols. For practical reasons, study participants, care providers and on-site investigators cannot be masked for investigational device versus comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of investigational device during sedation (Experimental): Intra-individual randomised paired crossover evaluation of airway patency with investigational device in volunteer study participants [I-II] and study patients [III-IV] at low, moderate and deep levels of steady-state sedation [I-II], and during procedural sedation according to SOC for scheduled colonoscopy [III] or ureteral catheterisation [IV].
  Interventions: Device: Investigational device [I-IV]
- Use of comparator during sedation (Active Comparator): Intra-individual randomised paired crossover evaluation of airway patency with comparator (biteblock [I-II] or no device [II-IV]) in volunteer study participants [I-II] and study patients [III-IV] at low, moderate and deep levels of steady-state sedation [I-II], and during procedural sedation according to SOC for scheduled colonoscopy [III] or ureteral catheterisation [IV].
  Interventions: Device: Comparator [I-IV]

INTERVENTIONS:
Device: Investigational device [I-IV] — Intra-individual randomised paired crossover evaluation of airway patency with investigational device in volunteer study participants [I-II] and study patients [III-IV] at low, moderate and deep steady-state sedation [I-II] or procedural sedation according to SOC [III-IV].
  Arms: Use of investigational device during sedation
Device: Comparator [I-IV] — Intra-individual randomised paired crossover evaluation of airway patency with comparator (biteblock [I-II] or no device [II-IV]) in volunteer study participants [I-II] and study patients [III-IV] at low, moderate and deep levels of steady-state sedation [I-II], and during procedural sedation according to SOC for scheduled colonoscopy [III] or ureteral catheterization [IV].
  Other Names: • Biteblock [I-II] • No device [II-IV]
  Arms: Use of comparator during sedation

SUMMARY:
The goal of this four-part preclinical [I-II] and clinical [III-IV] trial is to compare, with randomised crossover study design [I-IV], a new medical airway device with standard procedure (biteblock or no device) for upper airway patency during sedation with intravenous propofol [I-IV].

- Page 1 of 9 [DRAFT] - The two main questions it aims to answer are if this new airway device is superior to standard procedure with respect to

* maintenance of spontaneous ventilation [I] and upper airway volumes [II] at moderate and deep steady-state levels of sedation in healthy volunteer study participants, and
* fewer and less lasting bedside signs of respiratory depression [III-IV], and less adjuvant use of manual airway support [III-IV] during procedural sedation (PS) according to standard of care(SOC) in study patients scheduled for colonoscopy or ureteral catheterisation under PS. Owing to the crossover study design used throughout the trial, there are no comparison groups of study participants [I-II] or study patients [III-IV].

DETAILED DESCRIPTION:
OVERALL SYNOPSIS: I: Systematic evaluation, in supine body position, of O2 and ETCO2 monitoring at defined relevant levels of O2 supply by ID versus nasal cannula in non-sedated spontaneously breathing healthy volunteer study participants, and of respiratory function with ID versus biteblock during no, light (Ramsey levels 1-2), moderate (Ramsey level 3), and deep (Ramsey level 4) sedation with propofol in spontaneously breathing healthy volunteer study participants. Continuous supply of pure (instead of 30-35% according to SOC) O2 will at least three-fold the time until hypoxia may result from loss of airway patency during comparative evaluation of biteblock. II: Systematic evaluation, in supine body position, of MRI-derived anteroposterior transpharyngeal distances with ID versus biteblock or no device during no, light, moderate and deep sedation (as reported above) with propofol in spontaneously breathing healthy volunteer study participants. Continuous supply of pure (instead of 30-35% according to SOC) O2 will at least three-fold the time until hypoxia may result from loss of airway patency during comparative evaluation of biteblock and no device. III: Systematic evaluation in various body positions (as required by the procedural intervention) of the cumulative duration of adjuvant manual airway support (seconds), of perceived sedational comfort, sedational usability, and procedural conditions (VAS units), and of individual preference (ID or standard procedure if non-blinded; first or second intervention if blinded), with ID versus standard procedure (no device) during sedation according to SOC for scheduled colonoscopy in spontaneously breathing study patients. IV: Systematic evaluation in supine body position of the cumulative duration of adjuvant manual airway support (seconds), of perceived sedational comfort, sedational usability, and procedural conditions (VAS units), and of individual preference (ID or standard procedure if non-blinded; first or second intervention if blinded), with ID versus standard procedure (no device) during sedation according to SOC for scheduled ureteral catheterization in spontaneously breathing study patients. BACKGROUND: Procedural sedation (PS) is being increasingly used all over the world for diagnostic and therapeutic in- and out-hospital diagnostic and therapeutic interventions in various clinical settings. During PS, sedationists aim to reduce patient consciousness to levels enabling the procedure to be carried out smoothly with minimum intraprocedural discomfort, and with minimum fatigue and nausea in the early postprocedural period. However, collapse of soft tissue components in the upper airways at moderate and deep levels of sedation reduces or blocks airway flow, which may rapidly lead to hypoxia unless rapidly and appropriately managed at the bedside. According to a recent literature review, less severe respiratory adverse events during PS (bradypnoea, apnoea, mild hypoxia) often precede serious adverse respiratory events in clinical practice. However, medical devices currently used for airway patency during general anaesthesia all over the world, are not tolerated during light to moderate sedation, and hence cannot be used for airway patency during PS. By being well tolerated also in the awake state and during light sedation, the new investigational device (ID) for airway patency might hence increase patient safety, contribute to less stressful work environment, improve patient comfort, and contribute to more feasible, and hence more predictable, diagnostic and therapeutic procedures. The ID is expected to independently and reliably minimise the risk of partial or total airway obsruction - the main reason for sudden respiratory depression or even arrest - during PS. It may therefore enable the sedationist - inside or outside hospitals - to more readily and appropriately adapt the level of sedation to changing patient and procedural requirements without also having to take airway patency into continuous consideration. This prospective randomized paired crossover, single-centre trial in study participants will be carried out in four study parts [I-IV]. The two first preclinical parts [I-II] will include healthy female and male volunteer subjects to assess proof of concept, efficacy and safety of the ID at defined levels of sedation, and sedational comfort. The two later clinical parts [III-IV] will include female and male patients without serious medical comorbidity to further evaluate clinical safety in addition to sedational comfort, sedational usability, and procedural feasibility. Use of the ID will first be compared with standard procedure (biteblock [I-II] or no device [II]) with respect to maintenance of spontaneous breathing [I] or upper airway patency [II] at light, moderate and (particularly) deep levels of sedation in each study participant. NUMBER OF PARTICIPANTS: I. 12 (6 female) evaluable study participants (volunteer subjects). II. 12 (6 female) evaluable study participants (volunteer subjects). III. 16 (8 female) evaluable study participants (patients). IV. 16 (8 female) evaluable study participants (patients). DURATION: I-II: 2-3 weeks (February-March 2023). III-IV: 8-12 weeks (February-April 2023). PRIMARY OBJECTIVES: I: Comparison of tidal volumes assessed with modern ventilator equipment during light (Ramsey levels 1-2), moderate (Ramsey level 3) and deep (Ramsey level 4) sedation - achieved by estimated plasma levels of hypnotic drug (propofol) according to computerized infusion pump settings, and confirmed by bedside judgements according to Ramsey (levels 1-4), and by noninvasive bispectral index score (BIS) levels - during spontaneous breathing of pure oxygen in supine body position with ID versus biteblock. II: Comparison of anteroposterior transpharyngeal distances, determined by magnetic resonance imaging (MRI), during spontaneous breathing of pure oxygen at light, moderate, and deep sedation - achieved by estimated plasma levels of propofol according to computerized infusion pump settings, and assessed at the bedside according to Ramsey - in supine body position with ID versus biteblock, and versus no device. III: Comparison (by continuous observation and systematic recording) of cumulative duration of adjuvant use of manual airway support during sedation according to SOC, according to estimated plasma levels of propofol by computerized infusion pump settings, assessed at the bedside according to Ramsey (levels 1-4), for scheduled colonoscopy during spontaneous breathing in various body positions (as required by the procedure) with ID versus standard procedure (no device). IV: Comparison (by continuous observation and systematic recording) of cumulative duration of use of adjuvant manual airway support during sedation according to SOC, achieved and assessed as reported above and also by BIS levels, for scheduled ureteral catheterization during spontaneous breathing in supine body position with ID versus standard procedure (no device). SECONDARY OBJECTIVES: I: Evaluation of O2 and ETCO2 monitoring at defined levels of O2 supply by the ID versus by nasal cannula in non-sedated spontaneously breathing healthy volunteer study participants, and of respiratory rate, pressure and flow, and SpO2 levels, recorded with modern equipment for clinical routine supply and monitoring of general anaesthesia, at no, light (Ramsey levels 1-2), moderate (Ramsey level 3), and deep (Ramsey level 4) steady-state levels of sedation - achieved by algorithm-based estimated plasma levels of propofol according to computerized infusion pump settings, and assessed at the bedside according to Ramsey (levels 1-4), and by BIS levels, in healthy volunteer study participants in non-sedated spontaneously breathing healthy volunteer study participants spontaneous breathing pure O2 in the supine body position with ID versus standard procedure (biteblock). Survey evaluation of sedational comfort (VAS units). II: Survey evaluation of sedational comfort (VAS units). III-IV: Comparison of incidence (number) and duration (seconds) of interrupted ETCO2 monitoring, and of duration (second) and level (%) of hypoxia (SpO2 <95 %), during PS according to SOC, achieved and assessed as reported above, for scheduled colonoscopy [III] or ureteral catheterization [IV] during spontaneous breathing in various body positions as required by the procedural intervention [III] or in the supine body position [IV] with the ID versus standard procedure (no device). Survey evaluation of perceived sedational comfort (VAS units), and individual preference (ID or no device) by study participants (unblinded to interventional order), of perceived sedational usability (VAS units) and individual preference (ID or no device) by sedationists (unblinded to interventional order), and of perceived procedural conditions (VAS units) and individual preference (first or second study intervention) by procedural interventionists (blinded to interventional order) soon after completion of PS according to SOC with ID versus standard procedure (no device). PRIMARY STUDY ENDPOINT MEASURES: I: Absolute, and relative, differences in tidal volume (mL; mL/kg) between use of ID versus biteblock during deep (Ramsey level 4) sedation. II: Absolute, and relative, differences in anteroposterior transpharyngeal distances (mm and mm/kg, respectively) between use of ID versus biteblock or no device during deep (Ramsey level 4) sedation. III-IV: Absolute difference in cumulative duration of adjuvant manual airway support (seconds) between eight-minute use of ID versus eight-minute use of standard procedure (no device) during PS according to SOC for scheduled colonoscopy [III] or ureteral catheterization [IV]. SECONDARY STUDY ENDPOINT MEASURES: I: Endtidal concentrations of O2 and CO2 (%), and duration of interrupted tidal monitoring of O2 and CO2 (seconds), during defined relevant levels of O2 supply by the ID versus nasal cannula without sedation. Absolute, and relative, differences in tidal volume (mL; mL/kg) between ID and standard procedure (biteblock) during light (Ramsey levels 1-2) and moderate (Ramsey level 3) sedation. Differences in duration (seconds) of interrupted ETCO2 recording, in respiratory rate (min-1), in minimum and maximum airway pressures (cm H2O), in minimum and maximum absolute and relative airway flow (mL/min; mL/min/kg), and in SpO2 (%) during no, light (Ramsey levels 1-2), moderate (Ramsey level 3), and deep (Ramsey level 4) sedation. Individually perceived sedational comfort (VAS units). II: Absolute, and relative, differences in anterocrior transpharyngeal distance (mm; mm/kg) between use of ID versus standard procedure (biteblock or no device) during no, light (Ramsey levels 1-2) and moderate (Ramsey level 3) sedation. Individually perceived sedational comfort (VAS units). III-IV: Differences in cumulative duration (seconds) of interrupted ETCO2 monitoring, and of hypoxia (SpO2 <95 %), without adjuvant manual airway support, in perceived sedational comfort (VAS units), in perceived usability (VAS units), in perceived procedural conditions (VAS units), and in individual preference (ID or no device) by patient, sedationist and procedural interventionist during PS according to SOC with ID versus standard procedure (no device) for scheduled colonoscopy [III] or ureteral catheterization [IV].

ELIGIBILITY:
INCLUSION CRITERIA

Parts I-II:

Adult.

No known allergy or hypersensitivity to drugs used for routine sedation or to ID materials (polypropylene or ethylene vinylacetate).

Healthy with no medical comorbidity according to physician's judgement and physical examination.

No cognitive or psychosocial distress.

Complete or partial dentation.

No mobile teeth or reconstructions.

No orthodontic braces.

Non-pregnant.

Not breastfeeding.

Ability to communicate in Swedish.

No in situ magnetic device or implant [II].

Oral and written informed consent to inclusion as healthy volunteer study participant.

Parts III-IV:

Adult scheduled for elective colonoscopy [III] or ureteral catheterisation [IV] under procedural sedation with propofol.

No known allergy or hypersensitivity to drugs used for routine sedation or to ID materials (polypropylene or ethylene vinylacetate) in the ID.

Comorbidity ASA class I-III.

No cognitive or psychosocial distress.

Complete or partial dentation.

No mobile teeth or reconstructions.

No orthodontic braces.

Non-pregnant.

Not breastfeeding.

Ability to communicate in Swedish.

Oral and written informed consent to inclusion as study participant.

EXCLUSION CRITERIA

Parts I-IV:

Withdrawal of informed consent.

Suspected or manifest unforeseen allergic reaction.

Inability to obtain enough relevant study data for medical or technical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Difference in absolute and relative tidal volumes at deep sedation [I] | Estimated duration of measurements: 2-3 minutes per intervention. Estimated study period: 1-2 hours per participant.
  Nonblinded intra-individual randomised crossover evaluation, in a semi-closed-loop breathing system, of absolute (mL) and relative (mL/kg bodyweight) tidal volumes at deep steady-state level of propofol sedation between use of ID versus biteblock in supine spontaneously breathing adult volunteer study participants.
Difference in absolute and relative MRI-derived anteroposterior transpharyngeal distances at deep sedation [II] | Estimated duration of measurements: 2-3 min per intervention. Estimated study period: 1.5-2.5 h per participant.
  Nonblinded intra-individual randomised crossover evaluation, in an open breathing system, of absolute (mm) and relative (mm/kg bodyweight) anteroposterior transpharyngeal distances determined by MRI at deep steady-state level of propofol sedation between use of ID versus biteblock and versus no device in supine spontaneously breathing adult volunteer study participants.
Difference in adjuvant use of manual airway support during PS according to SOC [III-IV]. | Duration of measurements: 8 minutes per intervention. Estimated study period: 0.5-1 hours per patient.]
  Nonblinded intra-individual randomised crossover evaluation, in an open breathing system, of cumulative adjuvant use of manual airway support (seconds per minute) during PS with propofol according to SOC between use in spontaneously breathing adult volunteer study participants of ID versus no device in various body positions (as required by the interventional procedure) [III], or in supine body position [IV].

SECONDARY OUTCOMES:
Difference in absolute and relative tidal volumes at light and moderate sedation [I] | Estimated duration of measurements: 2-3 minutes per intervention. Estimated study period: 1-2 hours per participant.
  Nonblinded intra-individual randomised crossover evaluation, in a semi-closed-loop breathing system, of absolute (mL) and relative (mL/kg bodyweight) tidal volumes at moderate and at light steady-state levels of propofol sedation between use of ID versus biteblock in supine spontaneously breathing adult volunteer study participants.
Difference in duration (seconds) of maintained ETCO2 recording without sedation [I]. | Estimated duration of measurements: 2-3 min per intervention. Estimated study period: 1-2 h per participant.
  Nonblinded itra-individual randomised crossover evaluation, in an open breathing system, of duration (seconds per minute) of maintained ETCO2 recording at defined levels of O2 supply (1-2-3-5 L/min) between ID versus nasal cannula in supine spontaneously breathing awake adult volunteer study participants.
Difference in duration (seconds per minute) of hypoxia (SpO2 <95 %) during PS according to SOC [III-IV]. | Duration of measurements: 8 minutes per intervention. Estimated study period: 0.5-1 hours per patient.
  Nonblinded intra-individual randomised crossover evaluation, in an open breathing system, of duration (seconds per minute) of at least mild hypoxia (SpO2 <95 %) during PS according to SOC between ID versus no device in supine spontaneously breathing adult study patients.
Perceived sedational comfort [I-IV] and individual preference [III-IV] by study participants. | Estimated duration of data achievement: 3-4 minutes. Estimated study period: 0.5-2.5 hours per participant [I-IV].
  Nonblinded survey evaluation of perceived sedational comfort (VAS units) with ID in adult volunteer study participants subjected to light, moderate and deep steady-state levels of sedation [I-II], and in adult study patients subjected to PS according to SOC [III-IV], and of preference between ID and no device by adult study patients subjected to PS according to SOC [III-IV].
Perceived usability and individual preference by study sedationists [III-IV]. | Estimated duration of data achievement: 3-4 minutes. Estimated study period: 0.5-2.5 hours per participant [I-IV].
  Nonblinded individual survey evaluation in study sedationists of perceived usability of ID (preparation, induction, maintenance and emergence; VAS-units), and of individual preference, of ID versus no device, for PS according to SOC in adult study patients scheduled for elective colonoscopy [III] or ureteral catheterisation [IV].
Perceived procedural feasibility and individual preference by procedural interventionists [III-IV]. | Estimated duration of data achievement: 3-4 minutes. Estimated study period: 0.5-2.5 hours per participant [I-IV].
  Blinded individual survey evaluation in procedural interventionists of perceived procedural feasability of first versus second study intervention (ID or no device), and of individual preference, of first versus second study intervention, during PS according to SOC in adult study patients scheduled for elective colonoscopy [III] or ureteral catheterisation [IV].

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Åkeson, Professor, Principal Investigator — Lund University; Region Skane

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellin-Olsen J, Staender S. The Helsinki Declaration on Patient Safety in Anaesthesiology: the past, present and future. Curr Opin Anaesthesiol. 2014 Dec;27(6):630-4. doi: 10.1097/ACO.0000000000000131. PMID 25254572
- [Background] van Schaik EPC, Blankman P, Van Klei WA, Knape HJTA, Vaessen PHHB, Braithwaite SA, van Wolfswinkel L, Schellekens WM. Hypoxemia during procedural sedation in adult patients: a retrospective observational study. Can J Anaesth. 2021 Sep;68(9):1349-1357. doi: 10.1007/s12630-021-01992-6. Epub 2021 Apr 20. PMID 33880728
- [Background] Ciscar MA, Juan G, Martinez V, Ramon M, Lloret T, Minguez J, Armengot M, Marin J, Basterra J. Magnetic resonance imaging of the pharynx in OSA patients and healthy subjects. Eur Respir J. 2001 Jan;17(1):79-86. doi: 10.1183/09031936.01.17100790. PMID 11307760
- [Background] Youn AM, Ko YK, Kim YH. Anesthesia and sedation outside of the operating room. Korean J Anesthesiol. 2015 Aug;68(4):323-31. doi: 10.4097/kjae.2015.68.4.323. Epub 2015 Jul 28. PMID 26257843
- [Background] Roh WS, Kim DK, Jeon YH, Kim SH, Lee SC, Ko YK, Lee YC, Lee GH. Analysis of anesthesia-related medical disputes in the 2009-2014 period using the Korean Society of Anesthesiologists database. J Korean Med Sci. 2015 Feb;30(2):207-13. doi: 10.3346/jkms.2015.30.2.207. Epub 2015 Jan 21. PMID 25653494
- [Background] Muller M, Wehrmann T, Eckardt AJ. Prospective evaluation of the routine use of a nasopharyngeal airway (Wendl Tube) during endoscopic propofol-based sedation. Digestion. 2014;89(4):247-52. doi: 10.1159/000360000. Epub 2014 Jun 4. PMID 24903468
- [Background] Amornyotin S, Aanpreung P, Prakarnrattana U, Chalayonnavin W, Chatchawankitkul S, Srikureja W. Experience of intravenous sedation for pediatric gastrointestinal endoscopy in a large tertiary referral center in a developing country. Paediatr Anaesth. 2009 Aug;19(8):784-91. doi: 10.1111/j.1460-9592.2009.03063.x. PMID 19624366
- [Background] Cravero JP, Beach ML, Blike GT, Gallagher SM, Hertzog JH; Pediatric Sedation Research Consortium. The incidence and nature of adverse events during pediatric sedation/anesthesia with propofol for procedures outside the operating room: a report from the Pediatric Sedation Research Consortium. Anesth Analg. 2009 Mar;108(3):795-804. doi: 10.1213/ane.0b013e31818fc334. PMID 19224786
- [Background] Eastwood PR, Szollosi I, Platt PR, Hillman DR. Collapsibility of the upper airway during anesthesia with isoflurane. Anesthesiology. 2002 Oct;97(4):786-93. doi: 10.1097/00000542-200210000-00007. PMID 12357141
- [Result] Hinkelbein J, Lamperti M, Akeson J, Santos J, Costa J, De Robertis E, Longrois D, Novak-Jankovic V, Petrini F, Struys MMRF, Veyckemans F, Fuchs-Buder T, Fitzgerald R. European Society of Anaesthesiology and European Board of Anaesthesiology guidelines for procedural sedation and analgesia in adults. Eur J Anaesthesiol. 2018 Jan;35(1):6-24. doi: 10.1097/EJA.0000000000000683. PMID 28877145